CLINICAL TRIAL: NCT06073327
Title: Short-term Cocoa Supplementation Influences Long-chain n-3 Polyunsaturated Fatty Acid Concentration and Microbiota Composition in Elite Male Football Players
Brief Title: Short-term Cocoa Supplementation and Elite Soccer Players
Acronym: COCOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Padova_Soccer
Record Dates: First submitted 2023-06-01; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-05

CONDITIONS: Dyslipidemias; Fatty Acid; Metabolic Disorder
Keywords: fatty acid; soccer; dark chocolate
MeSH Terms: conditions — Dyslipidemias; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dark Chocolate (Experimental): Dark chocolate group was provided with 30g of dark chocolate (high in flavanol) for 30 days
  Interventions: Dietary Supplement: dark chocolate
- White Chocolate (Sham Comparator): White chocolate group was provided with30g of white chocolate (0 mg/g of polyphenol) for 30 days
  Interventions: Dietary Supplement: White chocolate

INTERVENTIONS:
Dietary Supplement: dark chocolate — 30g of dark or white chocolate was provided by the nutritionist for 30 days
  Arms: Dark Chocolate
Dietary Supplement: White chocolate — 30g of white chocolate was provided by the nutritionist for 30 days
  Arms: White Chocolate

SUMMARY:
The goal of this interventional study was to investigate the impact of daily ingestion of 30g of dark chocolate on omega-3 fatty acid status and gut microbial community in professional soccer players.

The main questions it aims to answer are:

Can 30g of dark chocolate positively influence the metabolism of polyunsaturated fatty acid (PUFAs) and, particularly, arachidonic acid (AA): eicosapentaenoic acid (EPA) ratio? Can 30g of dark chocolate change the microbial composition in professional soccer players? Elite male soccer players were randomly divided into 2 groups. One group was provided with 30g of dark chocolate 88% (2,5 mg/g of polyphenol) and one group, as control, was provided with with 30g of white chocolate (0 mg/g of polyphenol). Each group ingested the chocolate intervention as a "solid bar" in the morning (before 9:00 am) every day for 4 weeks. The dark chocolate and white chocolate were provided every morning to each subject by the nutritionist of each team, while, during off days, the chocolate was portioned into individual serving sizes and provided to each player. Adherence was checked by the nutritionist.

For each assessment, the participants arrived at the training center in the morning, after an overnight fast. Before the beginning and the end of the study, a 3-days food record (3dr) was recorded (2 weekdays and 1 week-end day) by the nutritionist. Blood was collected between 08:00 and 09:00 hours, fecal sample was delivered within the end of the morning, and anthropometry measures were determined.

DETAILED DESCRIPTION:
This study was conducted in May 2022. Elite male soccer players (n=38) were randomly divided into two groups. The dark chocolate group (DC N=19) was provided with 30g of dark chocolate 88% (Novi Nero Nero 88% cacao, Elah Dufour S.p.A., Strada Serravalle 73, Novi Ligure) (2,5 mg/g of polyphenol). The white chocolate group (WC n=19) was provided with 30g of white chocolate. (Bianco Novi, Elah Dufour S.p.A., Strada Serravalle 73, Novi Ligure) (0 mg/g of polyphenol). Each group ingested the chocolate intervention as a "solid bar" in the morning (before 9:00 am) every day for 4 weeks. The participants were instructed to refrain from consuming chocolate or flavanol-containing products (i.e., blueberry, strawberry, blackberry, green tea, red wine, and pomegranate juice), starting from 3 days before the beginning of the study and throughout the intervention period. The dark chocolate and white chocolate were provided every morning to each subject by the nutritionist of each team, while, during off days, the chocolate was portioned into individual serving sizes and provided to each player. Adherence was checked by the nutritionist.

For each assessment, participants arrived at the training center in the morning, after an overnight fast. Before the beginning and the end of the study, a 3-days food record (3DR) was recorded (2 weekdays and 1 week-end day) by the nutritionist, blood was collected between 08:00 and 09:00 hours, fecal sample was delivered within the end of the morning, and anthropometry measures were determined. Briefly, for stool samples, athletes were asked to collect their fecal material (single defecation) in a plastic vial and place the vial in a labelled box. The nutritionist and/or the doctor of each team immediately collected the fresh stool samples and delivered them within 72h to the research hub facility (University of Padova, Department of Biomedical Science).

ELIGIBILITY:
Inclusion Criteria:

• Elite football players playing in Serie A teams

Exclusion Criteria:

* Any disease or serious medical condition
* Probiotic use
* Special diet such as vegan or vegetarian or high-fiber
* Use of specific medications such as: non-steroidal anti-inflammatory drugs, antibiotics and statins taken in the last week

Ages: 18 Years to 38 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Plasmatic level of arachidonic acid and eicosapentaenoic acid (AA:EPA) ratio | 1 month
  Investigate the impact of daily ingestion of 30g of dark chocolate on omega-3 fatty acid status in professional soccer players
Main compositional changes in gut microbiota | 1 month
  Investigate the impact of daily ingestion of 30g of dark chocolate gut microbial community in professional soccer players

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- University of Padova, Padua, Italy